CLINICAL TRIAL: NCT01463358
Title: Prevention of Syncope by Cardiac Pacing in Patients With Bifascicular Block
Acronym: PRESS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GDT-20040601-PRESS-1
Record Dates: First submitted 2011-06-27; First posted 2011-11-01 (Estimated); Results first posted 2021-04-19 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-03

CONDITIONS: Bifascicular Block; Syncope
Keywords: Syncope; Bifascicular block; Bradycardia pacing
MeSH Terms: conditions — Syncope

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DDI30 (Other): Control group based only on backup pacing with lower rate 30 ppm
  Interventions: Device: DDD60 (INSIGNIA® pacing systems Guidant (Boston Scientific)
- DDD60 (Active Comparator): Treatment arm based on full pacing support (60 Lower Rate)
  Interventions: Device: DDD60 (INSIGNIA® pacing systems Guidant (Boston Scientific)

INTERVENTIONS:
Device: DDD60 (INSIGNIA® pacing systems Guidant (Boston Scientific) — pacing in DDD60 is supposed to prevent events of syncope, presyncope of cardioinhibitory origin and symptom associated to av block
  Other Names: INSIGNIA® pacing systems Guidant (Boston Scientific)
  Arms: DDD60
Device: DDD60 (INSIGNIA® pacing systems Guidant (Boston Scientific) — pacing in DDDI30 is supposed to act as a safety backup upfront to episodes of syncope, presyncope or AV block, but not supposed to reduce symptoms.
  Other Names: INSIGNIA® pacing systems Guidant (Boston Scientific)
  Arms: DDI30

SUMMARY:
Study Objective

The purpose of this study is to evaluate the efficacy of bradycardia pacing with respect to patient symptoms in patients with bifascicular block and syncope of unexplained origin.

DETAILED DESCRIPTION:
Primary endpoint

First occurrence of a composite of Syncope of any origin OR Presyncopal episode with documented cardioinhibitory origin OR Atrioventricular block of any degree; all associated with patient symptoms

Design:

* Randomized, prospective, single blinded, two parallel arms
* Treatment group : DDD60 - programmed in DDD mode / 60 lower limit
* Control Group: DDI30 - programmed in DDI mode / 30 lower limit
* Randomization type: block randomization: Block size: 4, allocation ratio 1:1

Sample: 100 patients

Population

* Patients with bifascicular block with at least one syncopal episode within the last 6 months preceding enrollment.
* Patients should be negative to a series of pre-enrollment screening in order to exclude:
* Brady-tachy syndrome, vasovagal syncope or carotid sinus syndrome, atrial fibrillation, inducible AV block
* Ejection fraction >=40%
* Mean nocturnal heart rate >=35 bpm

ELIGIBILITY:
Inclusion Criteria:

* Evidence of Bifascicular block
* At least one episode of syncope during last 6 months from the enrollment

Exclusion Criteria:

* Patients with Brady-tachy syndrome that needs of pacemaker to prevent the symptomatic bradycardia o symptomatic tachycardia arrhythmia
* Patients with vasovagal syndrome by positive TTT or carotid sinus syndrome
* Patients with Chronic Atrial Fibrillation
* Patients with Atrial Ventricular Block induces at EPS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2005-03; Primary Completion 2011-02 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Santini, MD,FESC,FACC, Principal Investigator — Ospedale San Filippo Neri, Roma, Italy
Locations (12):
- Italy (12):
  - Ospedale Santa Maria Annunziata, Bagno a Ripoli
  - Azienda Ospedaliera S. Sebastiano, Caserta
  - Ospedale Valduce, Como
  - Azienda Ospedaliera Osp. Maggiore, Crema
  - Nuovo Ospedale S. Giovanni di Dio, Florence
  - Ospedale Villa Scassi, Genova
  - Ospedale Umberto I, Mestre
  - Ospedale GB Grassi, Ostia - Roma
  - Ospedale Civile G. De Lellis, Rieti
  - Azienda Ospedaliera S. Filippo Neri, Roma
  - Ospedale Sandro Pertini, Roma
  - Policlinico Casilino, Roma

REFERENCES:
- [Derived] Brignole M, Donateo P, Tomaino M, Massa R, Iori M, Beiras X, Moya A, Kus T, Deharo JC, Giuli S, Gentili A, Sutton R; International Study on Syncope of Uncertain Etiology 3 (ISSUE-3) Investigators. Benefit of pacemaker therapy in patients with presumed neurally mediated syncope and documented asystole is greater when tilt test is negative: an analysis from the third International Study on Syncope of Uncertain Etiology (ISSUE-3). Circ Arrhythm Electrophysiol. 2014 Feb;7(1):10-6. doi: 10.1161/CIRCEP.113.001103. Epub 2013 Dec 12. PMID 24336948
- [Derived] Santini M, Castro A, Giada F, Ricci R, Inama G, Gaggioli G, Calo L, Orazi S, Viscusi M, Chiodi L, Bartoletti A, Foglia-Manzillo G, Ammirati F, Loricchio ML, Pedrinazzi C, Turreni F, Gasparini G, Accardi F, Raciti G, Raviele A. Prevention of syncope through permanent cardiac pacing in patients with bifascicular block and syncope of unexplained origin: the PRESS study. Circ Arrhythm Electrophysiol. 2013 Feb;6(1):101-7. doi: 10.1161/CIRCEP.112.975102. Epub 2013 Feb 6. PMID 23390123

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | DDI30 | DDD60
Started | 49 | 52
Completed | 46 | 47
Not Completed | 3 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DDI30 | DDD60 | Total
Number analyzed (Participants) | 49 | 52 | 101
Age, Continuous [Mean (Standard Deviation); unit: years] | 78 (8) | 77 (8) | 77 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 17 | 40
  Male | 26 | 35 | 61
Region of Enrollment [Number; unit: participants]
  Italy | 49 | 52 | 101

OUTCOME MEASURES:

1. Primary Outcome: Combined Endpoint Defined as First Occurrence Among the Following Events 1)Syncope Episode of Any Origin; 2)Presyncopal Episode With Documented Cardioinhibitory Origin 3) Atrioventricular Block of Any Degree Associated With Patient Symptoms
Description: Number of participants experiencing syncope episodes, symptomatic pre-syncopal episodes associated with a device intervention (ventricular pacing) and symptomatic episodes associated with documentation of intermittent or permanent atrio-ventricular block
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | DDI30 | DDD60
Number analyzed (Participants) | 49 | 52
Participants | 16 | 7

2. Secondary Outcome: Occurrence of First Symptomatic Episode (Syncope or Pre-syncope), Independently From Origin.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | DDI30 | DDD60
Number analyzed (Participants) | 49 | 52
Participants | 22 | 13

3. Secondary Outcome: Atrial Fibrillation
Description: patients presenting with at least one episode of atrial fibrillation during the 2 years follow up period
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | DDI30 | DDD60
Number analyzed (Participants) | 49 | 52
Participants | 9 | 18

ADVERSE EVENTS:
Time Frame: 2 years
Description: number of subjects with serious and non-serious adverse events of cardiac and non-cardiac origin, with identification of organ cause. Method for systematic assessment: regular investigator assessment at follow up.
Groups:
- DDI30: Control group based only on backup pacing with lower rate 30 ppm DDD60 (INSIGNIA® pacing systems Guidant (Boston Scientific): pacing in DDDI30 is supposed to act as a safety backup upfront to episodes of syncope, presyncope or AV block, but not supposed to reduce symptoms.
- DDD60: Treatment arm based on full pacing support (60 Lower Rate) DDD60 (INSIGNIA® pacing systems Guidant (Boston Scientific): pacing in DDD60 is supposed to prevent events of syncope, presyncope of cardioinhibitory origin and symptom associated to av block
Arm/Group | DDI30 | DDD60
All-Cause Mortality (participants affected / at risk) | 2/49 | 2/52
Serious Adverse Events (participants affected / at risk) | 33/49 | 23/52
Other Adverse Events (participants affected / at risk) | 22/49 | 20/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DDI30 (N=49) | DDD60 (N=52)
Syncope (Cardiac disorders) | 7 (9) | 7 (10)
atrio-ventricular block (Cardiac disorders) | 8 (9) | 2 (2)
symptomatic bradycardia (Cardiac disorders) | 9 (9) | 1 (1)
symptomatic atrial arrhyhtmias (Cardiac disorders) | 0 (0) | 2 (3) — serious: requiring hospitalizations
ventricular arrhyhtmias (Cardiac disorders) | 0 (0) | 1 (1)
Heart Failure exhacerbation (Cardiac disorders) | 2 (2) | 5 (5)
Miocardial Infarction (Cardiac disorders) | 0 (0) | 1 (1)
intervention for coronary artery disease (Cardiac disorders) | 2 (2) | 0 (0) — Coronary artery Bypass Graft or Percutaneous angioplasty
Stroke (Cardiac disorders) | 1 (1) | 0 (0)
transient ischemic attack (Cardiac disorders) | 1 (1) | 0 (0)
peripheral vascular disease (Vascular disorders) | 1 (1) | 0 (0)
Vascular encephalopathy (Vascular disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (COPD) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3)
Loss of pacemaker capture (Product Issues) | 3 (3) | 0 (0) — requiring invasive system revision
Pacing lead dislodgment (Product Issues) | 1 (1) | 1 (1) — requiring invasive system revision
Pacemaker system infection (Product Issues) | 2 (2) | 1 (1)
Gastrointestinal disease (Gastrointestinal disorders) | 0 (0) | 2 (2)
Musculoskeletal trauma (Musculoskeletal and connective tissue disorders) | 5 (5) | 2 (2)
Renal disease (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary disease (Renal and urinary disorders) | 1 (1) | 1 (1)
Fever/virus (General disorders) | 0 (0) | 1 (1)
Tumor (General disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DDI30 (N=49) | DDD60 (N=52)
Dizziness (Cardiac disorders) | 15 (23) | 8 (8)
symptomatic Atrial Arrhythmias (Cardiac disorders) | 0 (0) | 2 (2) — non-serious: not requiring hospitalisation
Heart Failure (Cardiac disorders) | 5 (6) | 4 (4) — non-serious: treated with variation to medical therapy
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
pacemaker signal oversensing/undersensing (Product Issues) | 6 (7) | 9 (14) — non serious: resolved with pacemaker reprogramming
pacemaker: rise in pacing threshold (Product Issues) | 2 (2) | 3 (3) — non serious: resolved with pacemaker reprogramming

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No